CLINICAL TRIAL: NCT01224652
Title: A Randomized, Multicenter Phase III Study to Assess the Efficacy of Paclitaxel Versus Irinotecan in Patients With Recurrent or Metastatic Gastric Cancer Who Progress Following First-line Therapy
Brief Title: Efficacy Study of Paclitaxel Versus Irinotecan in Patients With Recurrent or Metastatic Gastric Cancer Who Progress Following First-line Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Cancer Study Group (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Tae-You Kim, Chairperson of Stomach Cancer Committee, Korean Cancer Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-ST10-01
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; paclitaxel; irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paclitaxel (Experimental): Paclitaxel 70 mg/m2 on Days 1, 8 and 15 of a 28-day cycle
  Interventions: Drug: Paclitaxel
- irinotecan (Experimental): irinotecan 150 mg/m2 on Days 1 and 15 of a 28-day cycle
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel, 70 mg/m2 will be administered as an intravenous (IV) infusion over 1 hour on Days 1, 8 and 15 of a 28-day cycle
  Arms: paclitaxel
Drug: Irinotecan — irinotecan 150 mg/m2 will be administered as an intravenous (IV) infusion over 1 hour on Days 1 and 15 of a 28-day cycle
  Arms: irinotecan

SUMMARY:
The primary objectives of this study is to compare the efficacy of paclitaxel monotherapy with irinotecan monotherapy as defined by progression-free survival (PFS), in all patients with recurrent and metastatic gastric cancer who progress following first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric adenocarcinoma in tissue/cell
* Recurrent or metastatic gastric cancer that has progressed following first- line therapy
* Patients must be ≥18 years of age.
* ECOG performance status ≤ 2
* At least one lesion (measurable or non-measurable but evaluable) according to RECIST criteria
* Normal organ and bone marrow function measured within 2 weeks prior to administration of study treatment as defined below: Haemoglobin ≥ 9.0 g/dL White blood cells (WBC) ≥ 3000/µL Absolute neutrophil count (ANC) ≥ 1500/µL Platelet count ≥ 100 x 103/µL Total bilirubin ≤ 1.5 x upper normal limit (UNL) Creatinine clearance ≥ 60 ml/min or Serum creatinine ≤ 1.5 x UNL AST (SGOT)/ALT (SGPT) ≤ 2.5 x UNL unless liver metastases are present in which case it must be ≤ 5x UNL
* Life expectancy ≥ 12 weeks.
* Written informed consent
* Provision of informed consent for genetic research (In case of optional genetic research)

Exclusion Criteria:

* More than one prior chemotherapy regimen for the treatment of gastric cancer in the metastatic or recurrent setting.
* Treatment with any investigational product during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
* Any previous treatment with a taxane, including paclitaxel and docetaxel or irinotecan, in the metastatic or recurrent setting.
* Patients with second primary cancer, except: adequately treated non- melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥5 years.
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used).
* Ongoing toxicities (>CTCAE grade 2) caused by previous cancer therapy.
* Clinically proven gastric outlet obstruction or CTCAE grade 3 or grade 4 upper GI bleeding
* Medically uncontrolled, clinically significant heart disease or infection
* Patients with symptomatic uncontrolled brain metastases.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Women who have pregnancy potential or willing to pregnant. Pregnant and breastfeeding women.
* Others Poor medical risk due to a serious, uncontrolled medical disorder, non- malignant systemic disease or active, uncontrolled infection Any psychiatric disorder that prohibits obtaining informed consent and regular follow-up. Inappropriate patient for subjects of this study on investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | every 8 weeks
  Tumor evaluation using RECIST v1.1

SECONDARY OUTCOMES:
Safety | up to 4 weeks after last administration of chemotherapy
  Number of Participants and toxicity grade accordong to NCI-CTCAE v3.0 as a Measure of Safety
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tae-You Kim, M.D., Ph.D., Study Chair — Korean Cancer Stusy Group stomach Cancer Committee
Locations (2):
- South Korea (2):
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee KW, Maeng CH, Kim TY, Zang DY, Kim YH, Hwang IG, Oh SC, Chung JS, Song HS, Kim JW, Jeong SJ, Cho JY. A Phase III Study to Compare the Efficacy and Safety of Paclitaxel Versus Irinotecan in Patients with Metastatic or Recurrent Gastric Cancer Who Failed in First-line Therapy (KCSG ST10-01). Oncologist. 2019 Jan;24(1):18-e24. doi: 10.1634/theoncologist.2018-0142. Epub 2018 Aug 20. PMID 30126861